CLINICAL TRIAL: NCT05693207
Title: EMG to Detect and Monitor Freezing of Gait Among People With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-21-NG-0515-CTIL
Record Dates: First submitted 2022-12-27; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2022-11

CONDITIONS: Evaluation of Muscle Contraction in People With PD

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- People with iPD with freezing of gait (Experimental)
  Interventions: Device: EMG
- People with iPD without freezing of gait (Other): control group
  Interventions: Device: EMG

INTERVENTIONS:
Device: EMG — wearables EMG
  Other Names: Accelerometers and gyroscopes

SUMMARY:
The main goal of this study is to evaluate, via EMG (electromyography) system, the muscle activity in the lower limbs, to understand the contribution of the muscle activity to FOG (freezing of gait) in Parkinson's patients. The phenomenon of FOG appears in advanced cases of Parkinson's disease (PD) and can lead to an increased risk of falls. There are several approaches claiming that there is abnormal activity in the calf muscles and the freezing events in Parkinson's patients. In the clinic, monitoring FOG is done subjectively, usually through observations or through questionnaires. As a result, the information about the phenomenon may be biased and insensitive. With an electromyographic monitor (EMG), objective information about the muscular activity during normal walking and during unusual events can be obtained.

DETAILED DESCRIPTION:
The subject will arrive independently at the Tel Aviv Medical Center. After explaining the course of the study and signing a consent form, the subject will be administered the MoCA questionnaire to assess the cognitive state.

During this session, the patient will undergo gait evaluation using motion sensors and an EMG device.

This meeting will last up to an hour, according to the following breakdown:

Explanation of the test (10 min) Preparing the skin (light disinfection with alcohol) for EMG adhesion (10 min.) Performing of the test (20 minutes) Summary and discharge (5 min).

ELIGIBILITY:
Inclusion criteria for patients:

1. Men and women aged 40-89.
2. Patients with idiopathic Parkinson's disease according to the diagnosis of a neurologist, who are able to walk with or without a walking aid for at least 5 minutes.
3. 21 or above in MoCA test.
4. people who gave their written and oral consent to participate in the study.

Inclusion criteria for healthy people:

1. Men and women aged 40-89.
2. 24 or above in MoCA test.
3. Without a neurological, cardiovascular or orthopedic disorder, which could affect the normal walking pattern, and all within the researcher's decision.

Criteria for exclusion from the experiment:

1. The patient has serious side effects that are not suitable for continuing in the study.
2. The patient does not wish to continue his participation in the study.

Exclusion criteria for Parkinson's patients:

1. Neurological or other psychiatric disorder (such as MSA, PSP, after a stroke with neurological signs, dementia diseases, clinical depression) at the researcher's decision.
2. History of head injury - traumatic brain injury or cerebrovascular accident (CVA)
3. This study will not include pregnant women and children.

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-07 (Actual); Primary Completion 2023-05-23 (Estimated); Study Completion 2023-12-23 (Estimated)

PRIMARY OUTCOMES:
Percentage time of co-contractions | 60 minutes
  The time of co-contraction during walking will be higher among people with FOG.

CONTACTS AND LOCATIONS:
Overall Officials: Nir Giladi, Prof, Principal Investigator — Study Principal Investigator Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel aviv medical center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pringsheim T, Jette N, Frolkis A, Steeves TD. The prevalence of Parkinson's disease: a systematic review and meta-analysis. Mov Disord. 2014 Nov;29(13):1583-90. doi: 10.1002/mds.25945. Epub 2014 Jun 28. PMID 24976103
- [Background] Bloem BR, Hausdorff JM, Visser JE, Giladi N. Falls and freezing of gait in Parkinson's disease: a review of two interconnected, episodic phenomena. Mov Disord. 2004 Aug;19(8):871-84. doi: 10.1002/mds.20115. PMID 15300651
- [Background] Silva de Lima AL, Evers LJW, Hahn T, Bataille L, Hamilton JL, Little MA, Okuma Y, Bloem BR, Faber MJ. Freezing of gait and fall detection in Parkinson's disease using wearable sensors: a systematic review. J Neurol. 2017 Aug;264(8):1642-1654. doi: 10.1007/s00415-017-8424-0. Epub 2017 Mar 1. PMID 28251357
- [Background] Hanein Y, Mirelman A. The Home-Based Sleep Laboratory. J Parkinsons Dis. 2021;11(s1):S71-S76. doi: 10.3233/JPD-202412. PMID 33682729
- [Background] Inzelberg L, David-Pur M, Gur E, Hanein Y. Multi-channel electromyography-based mapping of spontaneous smiles. J Neural Eng. 2020 Apr 9;17(2):026025. doi: 10.1088/1741-2552/ab7c18. PMID 32271717
- [Background] Mazzetta I, Zampogna A, Suppa A, Gumiero A, Pessione M, Irrera F. Wearable Sensors System for an Improved Analysis of Freezing of Gait in Parkinson's Disease Using Electromyography and Inertial Signals. Sensors (Basel). 2019 Feb 23;19(4):948. doi: 10.3390/s19040948. PMID 30813411